CLINICAL TRIAL: NCT07164703
Title: Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Brief Title: A Real-World Study of Precision Treatment for Advanced Cholangiocarcinoma Based on Molecular Subtyping
Status: Not yet recruiting | Type: Observational
Sponsor: Mao-Lin Yan (Other)
Responsible Party: Sponsor-Investigator, Mao-Lin Yan, Principal Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: FJPH-CCA-PT-2025; FJPH-CCA-PT-2025 (Other: Fujian Provincial Hospital)
Record Dates: First submitted 2025-08-31; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cholangiocarcinoma (Part 1)
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Precision Treatment Based on Molecular Subtyping (or Gene Mutations)
  Interventions: Drug: Targeted drugs or immunotherapies for cholangiocarcinoma based on targetable gene mutations.

INTERVENTIONS:
Drug: Targeted drugs or immunotherapies for cholangiocarcinoma based on targetable gene mutations. — Targeted drugs or immunotherapies for cholangiocarcinoma based on targetable gene mutations.

SUMMARY:
This is a multi-center, real-world study aiming to evaluate the efficacy and safety of precision treatment for advanced cholangiocarcinoma (CCA) with different molecular subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Histologically confirmed, unresectable advanced biliary tract carcinoma, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder cancer (diagnosed according to the 2025 Chinese Society of Clinical Oncology (CSCO) Guidelines for Biliary Tract Malignancies and confirmed by a multidisciplinary team). Must have a documented targetable gene mutation, including but not limited to: Fibroblast Growth Factor Receptor 2 (FGFR2) fusion/rearrangement, Isocitrate Dehydrogenase (NADP(+)) 1 (IDH-1) and Isocitrate Dehydrogenase (NADP(+)) 2 (IDH-2) mutations, Erb-B2 Receptor Tyrosine Kinase 2 (ERBB2/HER2) amplification and/or overexpression, B-Raf Proto-Oncogene, Serine/Threonine Kinase (BRAF) V600E mutation, Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) mutation, Neurotrophic Tyrosine Receptor Kinase (NTRK) fusion, Rearranged during Transfection (RET) fusion, Ring Finger Protein 43 (RNF43) mutation, MET Proto-Oncogene, Receptor Tyrosine Kinase (MET) amplification, Epidermal Growth Factor Receptor (EGFR) mutation, Phosphatidylinositol-4,5-Bisphosphate 3-Kinase Catalytic Subunit Alpha (PIK3CA) mutation, BRCA1 DNA Repair Associated (BRCA1)/BRCA2 DNA Repair Associated (BRCA2) mutation, Partner and Localizer of BRCA2 (PALB2) mutation, Vascular Endothelial Growth Factor Receptor (VEGFR) mutation, deficient Mismatch Repair (dMMR)/Microsatellite Instability-High (MSI-H), or Neuregulin 1 (NRG1) mutation.
3. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (measurable lesion defined as longest diameter ≥10 mm on Computed Tomography (CT)/Magnetic Resonance Imaging (MRI) scan).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Child-Pugh class A or B liver function. For patients with obstructive jaundice, total bilirubin must be ≤ 50 µmol/L. Biliary drainage is recommended if total bilirubin is > 50 µmol/L.
6. Adequate hematologic function: Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L, Hemoglobin (Hb) ≥ 8.5 g/L, Platelets (PLT) ≥ 75 × 10^9/L.
7. No history of severe arrhythmia or heart failure; no severe ventilation dysfunction or severe pulmonary infection; no acute or chronic renal failure with creatinine clearance > 40 mL/min.
8. Life expectancy of more than 3 months.

Exclusion Criteria:

1. Major surgery within 28 days prior to enrollment.
2. Presence of any unresolved toxicity of Grade ≥ 2 (according to Common Terminology Criteria for Adverse Events [CTCAE] v4.0) from prior anticancer therapy at the time of enrollment, with the exception of alopecia or Grade 2 anemia.
3. Known hypersensitivity to any components or excipients of the study drugs.
4. Presence of any active autoimmune disease or a history of autoimmune disease with an expected recurrence. Patients currently receiving immunosuppressants or systemic corticosteroids for immunosuppressive purposes.
5. Presence of other concurrent malignancies.
6. Presence of brain metastases or spinal cord compression.
7. Presence of any severe and/or unstable pre-existing medical conditions, mental illness, or other conditions that could compromise patient safety, the ability to provide informed consent, or adherence to the study procedures.
8. Pregnant or breastfeeding women.
9. History of organ transplantation.
10. Patients with proteinuria ≥ 1+ on urinalysis must undergo a 24-hour urine protein test. Patients with a 24-hour urine protein level ≥ 1g are excluded.
11. Clinically significant corneal or retinal disease confirmed by ophthalmologic examination.
12. Liver tumor burden exceeding 50%.
13. Hypothyroidism or hyperthyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female adults aged 18 to 75 years. Participants must have histologically confirmed, unresectable advanced biliary tract carcinoma, which encompasses intrahepatic or extrahepatic cholangiocarcinoma (CCA) and gallbladder cancer.A key criterion for inclusion is the presence of a documented targetable gene mutation, such as FGFR2 fusion/rearrangement, IDH-1 or IDH-2 mutations, ERBB2 (HER2) amplification/overexpression, BRAF V600E mutation, or others.Eligible patients are required to have at least one measurable lesion according to RECIST 1.1 criteria and a good performance status, indicated by an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1. Furthermore, participants must have a life expectancy of more than 3 months and adequate organ function, including Child-Pugh class A or B liver function and specified levels of hematologic and renal function.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | Four weeks after the initiation of medication
  The Objective response rate (ORR) was defined as the complete response (CR) rate or the partial response (PR) rate according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

SECONDARY OUTCOMES:
Overall survival, OS | From date of enrollment until the date of death from any cause, assessed up to 48 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Progression-free survival, PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
Disease control rate, DCR | Four weeks after the initiation of medication
  The Disease control rate (DCR) was defined as the complete response (CR) rate or the partial response (PR) rate or stable disease (SD) rate according to RECIST v1.1 criteria.
Treatment-related adverse events, TRAEs treatment-related adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 48 months
  The incidence, spectrum and severity of adverse events (AE) and serious adverse events (SAE) were determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) V5.0 standard. Dose suspension rate and dose termination rate due to adverse events.
Conversion Resection Rate, CRR | Four weeks after the initiation of medication until the day before surgery
  The proportion of all enrolled patients who meet the criteria for resectability and undergo surgical resection after receiving study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maolin Lin, Doctor, Study Chair — Department of Hepatobiliary and Pancreatic Surgery, Affiliated Provincial Hospital of Fuzhou University
Locations (1):
- Affiliated Provincial Hospital of Fuzhou University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No